CLINICAL TRIAL: NCT04233723
Title: Effect of Severe Trauma on Programmed Death Molecule (PD1) and Its Legend (PD1/L1) on T Lymphocytes and Correlation With Mortality
Brief Title: Effect of Severe Trauma on PD1 and Its Legend (PD1/L1) on T Lymphocytes and Correlation With Mortality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RRHennis, principal investigator, Assiut University
Other Study IDs: IRB171000017
Record Dates: First submitted 2019-03-15; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-02

CONDITIONS: Trauma Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — peripheral venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: peripheral blood samples — venous puncture

SUMMARY:
Unlike neuro-endocrine response to trauma; posttraumatic immune alterations are not easily carried out at bedside. The majority of trials were conducted in the intensive care usually hours to days post injury.

In this trial the investigators sought assess the immune responses during emergency department trauma resuscitation by looking at the biomarkers of severe injury by comparing T lymphocytes and programmed cell death molecules and its relation with mortality.

DETAILED DESCRIPTION:
Trauma is a major healthcare problem with a high mortality rate that might be caused by immune-suppression.

Trauma initiates an immunosuppressive response which is contributor tocell damage and could be a marker of multi organ failure and mortality.

Programmed cell death receptor-1 (PD-1) and programmed cell death receptor ligand-1 (PD-L1), which are co-inhibitory receptor molecules, may participate in trauma-induced immune-suppression.

Both sterile and infected trauma induce the systemic inflammatory response syndrome (SIRS), originally defined by pyrexia, tachycardia, hyperventilation and neutrophilia, the latter responding poorly to pathogens. (10) Accompanying these changes is a decrease in circulating basophil, eosinophil and natural killer precursors, which further weakens systemic immunity.

Apoptosis (Programmed Cell Death):

Programmed cell-death (PCD) is death of a cell in any form, mediated by an intracellular program. PCD is carried out in a regulated process, which usually confers advantage during an organism's life-cycle. Apoptosis and autophagy are both forms of PCD, but necrosis is a non-physiological process that occurs as a result of infection or injury.

Programmed cell death protein 1 Programmed cell death protein 1, also known as PD-1 and CD 279 (cluster of differentiation 279), is a protein that in humans is encoded by the PDCD1 gene. PD-1 is a cell surface receptor that belongs to the immunoglobulin super family and is expressed on T cells and pro-B cells. PD-1 binds two ligands, PD-L1 and PD-L2. PD-1, functioning as an immune checkpoint, plays an important role in down regulating the immune system by preventing the activation of T-cells, which in turn reduces autoimmunity and promotes self-tolerance.

Ligands PD-1 has two ligands, PD-L1 and PD-L2, which are members of the B7 family. Several lines of evidence suggest that PD-1 and its ligands negatively regulate immune responses PD-1 knockout mice have been shown to develop lupus-like glomerulo-nephritis and dilated cardiomyopathy Triggering PD-1, expressed on monocytes and up-regulated upon monocytes activation, by its ligand PD-L1 induces IL-10 production which inhibits CD4 T-cell function.

ELIGIBILITY:
Inclusion Criteria:

1. Adult trauma patients with blunt or penetrating injury.
2. Major injury:

   * Injury severity score > 15
   * Drop in hematocrit > 10 points
   * Transfusion of more than 6-10 units of packed RBCs
   * Serum lactate > 3 mmol/L
3. Mean arterial blood pressure ≤ 60 mmHg and/or systolic arterial blood pressure ≤ 90 mmHg.
4. Patients admitted to the ED within 6 hours after the onset of trauma

Exclusion Criteria:

- 1. age less than 18 years; 2. patients who died within 2 days of the onset of trauma; 3. patients who declined to consent; 4. Known pregnancy. 5. Patients with limb ischemia or peripheral vascular occlusion. 6. Patients admitted to the emergency trauma department after 6 hours of the trauma event.

7. Preexisting conditions as severe cardiovascular disease, uncontrolled hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: trauma emergency department and Trauma ICU of Assiut university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Measuring standard deviations of biomarkers of severe injury by comparing T lymphocytes and programmed cell death molecules and its relation with mortality. | 48 hours
  Results for normally distributed continuous variables will be expressed as mean value, standard deviation and inter-quartile range. Categorical data and dichotomous variables will be shown as number and percentage.
  Comparisons of continuous variables will be performed using independent t-test. Proportions will be compared with chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Ramy R Hennis, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engelberg-Kulka H, Amitai S, Kolodkin-Gal I, Hazan R. Bacterial programmed cell death and multicellular behavior in bacteria. PLoS Genet. 2006 Oct;2(10):e135. doi: 10.1371/journal.pgen.0020135. PMID 17069462
- [Background] Islam N, Whitehouse M, Mehendale S, Hall M, Tierney J, O'Connell E, Blom A, Bannister G, Hinde J, Ceredig R, Bradley BA. Post-traumatic immunosuppression is reversed by anti-coagulated salvaged blood transfusion: deductions from studying immune status after knee arthroplasty. Clin Exp Immunol. 2014 Aug;177(2):509-20. doi: 10.1111/cei.12351. PMID 24749651
- [Background] Murray CK, Hinkle MK, Yun HC. History of infections associated with combat-related injuries. J Trauma. 2008 Mar;64(3 Suppl):S221-31. doi: 10.1097/TA.0b013e318163c40b. PMID 18316966
- [Background] Kaczmarek A, Vandenabeele P, Krysko DV. Necroptosis: the release of damage-associated molecular patterns and its physiological relevance. Immunity. 2013 Feb 21;38(2):209-23. doi: 10.1016/j.immuni.2013.02.003. PMID 23438821